CLINICAL TRIAL: NCT02586181
Title: Effect of 1 Year Vitamin D or D Plus B-vitamins on Bone Markers in Elderly People
Brief Title: Effect of 1 Year Vitamin D or D Plus B-vitamins on Bone Markers in Elderly People (KnoVIB)
Acronym: KnoVIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Rima Obeid, Prof. (apl.) Dr., Universität des Saarlandes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Vitamins and bone markers
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Nutritional Supplement Toxicity
MeSH Terms: interventions — Vitamin D; Calcium; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D and Calcium (Placebo Comparator): a combination of dietary supplement including "all" 1200 IE Vitamin D3 plus 800 mg Calcium Carbonate
  Interventions: Dietary Supplement: Vitamin D and Calcium
- Vitamin D, Calcium, Vitamins B9, B6, B12 (Experimental): a combination of dietary supplement including "all" 1200 IE Vitamin D3 plus 800 mg Calcium Carbonate plus 0,5mg Folic acid, 50 mg B6, 0,5 mg B12
  Interventions: Dietary Supplement: Vitamin D, Calcium, Vitamins B9, B6, B12

INTERVENTIONS:
Dietary Supplement: Vitamin D and Calcium — a combination of dietary supplement including "all" 1200 IE Vitamin D3 plus 800 mg Calcium Carbonate
  1200 IE Vitamin D3 plus 800 mg Calcium Carbonate
  Arm: Experimental: Vitamin D, Calcium, Vitamins B9, B6, B12
  1200 IE Vitamin D3 plus 800 mg Calcium Carbonate plus 0,5mg Folic acid, 50 mg B6, 0,5 mg B12
  Arms: Vitamin D and Calcium
Dietary Supplement: Vitamin D, Calcium, Vitamins B9, B6, B12 — a combination of dietary supplement including "all" 1200 IE Vitamin D3 plus 800 mg Calcium Carbonate plus 0,5mg Folic acid, 50 mg B6, 0,5 mg B12
  Arms: Vitamin D, Calcium, Vitamins B9, B6, B12

SUMMARY:
The standard recommendation to prevent osteoporosis is to supplement low doses of vitamin D and calcium. Hyperhomocysteinemia has been related to increased risk of osteoporosis.

DETAILED DESCRIPTION:
The current study aimed at investigating if homocysteine-lowering effect (low doses of B-vitamins) will add any measurable beneficial effect on bone markers when added to the standard recommendations for prevention of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* age> 50 years,
* male and female

Exclusion Criteria:

* renal dysfunction,
* recent stroke or coronary event within the last 3 months,
* current cancer,
* antifolate treatment,
* ileum resection,
* existing B vitamins supplementation,
* megaloblastic anemia,
* osteoporotic patients treated with pharmacological doses of vitamin D or antiosteoporotic drugs.

Termination criteria were:

* indication for a high-dose vitamin B supplementation,
* coronary or vascular event,
* or surgical procedures during the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in bone formation markers | baseline, 6 and 12 months
  Concentrations of bone formation markers in plasma [OC (ng/ml), BAP (U/L)]: are measured: if all are increased indicate enhanced bone formation

SECONDARY OUTCOMES:
Changes in plasma choline and betaine | baseline and aftter 12 months
  plasma choline and betaine (all µmol/L): if both increased indicate saving betaine and choline
Changes in global DNA methylation | baseline and after 12 months
  global DNA methylation [line 1-methylation (expressed as %)]
Changes in gene-specific gene methylation | baseline and after 12 months
  After isolating DNA from whole blood, changes in methylation of targeted genes is studied (expressed as %)
Changes in TMAO | baseline and after 6 and 12 months
  Plasma concentrations of TMAO ((µmol/L) is measured
Changes in phospholipid concentration in plasma | baseline and after 12 months
  Plasma phospholipids ((µmol/L) are measured
Changes in concentrations of bone resorption markers | baseline, 6 and 12 months
  concentrations of bone resorption markers [plasma TRAP5b (U/L), urine DPD (nmol//mmol creatinine)]: if both are increased indicate enhanced bone resorption
Changes in plasma homocysteine concentrations | baseline, 6 and 12 months
  changes in plasma homocysteine (µmol/L) between the time points
Changes in plasma levels of folate | baseline, 6 and 12 months
  changes in serum and whole blood folate (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Rima Obeid, PhD, Principal Investigator — Universität des Saarlandes
Locations (1):
- University of Saarland, Homburg, Saarland, Germany

REFERENCES:
- [Result] Kirsch SH, Herrmann W, Kruse V, Eckert R, Graber S, Geisel J, Obeid R. One year B-vitamins increases serum and whole blood folate forms and lowers plasma homocysteine in older Germans. Clin Chem Lab Med. 2015 Feb;53(3):445-52. doi: 10.1515/cclm-2014-0540. PMID 25283139
- [Result] Hubner U, Geisel J, Kirsch SH, Kruse V, Bodis M, Klein C, Herrmann W, Obeid R. Effect of 1 year B and D vitamin supplementation on LINE-1 repetitive element methylation in older subjects. Clin Chem Lab Med. 2013 Mar 1;51(3):649-55. doi: 10.1515/cclm-2012-0624. PMID 23314556
- [Result] Herrmann W, Kirsch SH, Kruse V, Eckert R, Graber S, Geisel J, Obeid R. One year B and D vitamins supplementation improves metabolic bone markers. Clin Chem Lab Med. 2013 Mar 1;51(3):639-47. doi: 10.1515/cclm-2012-0599. PMID 23183751
- [Derived] Obeid R, Hubner U, Bodis M, Graeber S, Geisel J. Effect of adding B-vitamins to vitamin D and calcium supplementation on CpG methylation of epigenetic aging markers. Nutr Metab Cardiovasc Dis. 2018 Apr;28(4):411-417. doi: 10.1016/j.numecd.2017.12.006. Epub 2017 Dec 29. PMID 29395637
- [Derived] Obeid R, Awwad HM, Rabagny Y, Graeber S, Herrmann W, Geisel J. Plasma trimethylamine N-oxide concentration is associated with choline, phospholipids, and methyl metabolism. Am J Clin Nutr. 2016 Mar;103(3):703-11. doi: 10.3945/ajcn.115.121269. Epub 2016 Feb 10. PMID 26864355